CLINICAL TRIAL: NCT02223078
Title: Phase II, Randomised, Double-blind, Placebo-controlled, Parallel Group, Two Centre Study to Determine the Effect of G17DT on Plasma Gastrin Levels in Patients With Colorectal Cancer.
Brief Title: Two Center Study to Determine Effect of G17DT on Plasma Gastrin Levels in Patients With Colorectal Cancer.
Acronym: CC4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CC4
Record Dates: First submitted 2014-07-02; First posted 2014-08-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2014-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- G17DT (Experimental): Three 250 µg injections over a six week period (weeks 0,2 and 6)
  Interventions: Biological: G17DT
- Placebo (Placebo Comparator): Three 250 µg injections of a placebo over a six week period (weeks 0,2 and 6)
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: G17DT
  Arms: G17DT
Biological: Placebo Comparator
  Arms: Placebo

SUMMARY:
Pancreatic, gastric, and colorectal cancers have all been shown to overexpress the gastrin gene and to be sensitive to the trophic effects of the gastrin in animal models. The hypothesis of this study is that G17DT will elicit specific and high-affinity antibodies that will bind gastrin-17, thus preventing the trophic activity of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed colorectal carcinoma for whom no other anti-cancer treatment was anticipated during the three month period of study.
* Patients taking a proton pump inhibitor at a fixed daily dose which had remained unchanged for at least six weeks preceding screening and was not anticipated to change during the study.
* Proton pump inhibitor compliance of ~70% (to be measured between screening and baseline (week 0)).
* Male or female patients from 18 to 65 years of age.
* Patients with a life expectancy of over three months.
* World Health Organisation (WHO) Performance Status of 0 to 1.
* Written informed consent given.

Exclusion Criteria:

* Patients in receipt of histamine H2-receptor (H2 receptor) antagonists or any other antacid therapy, other than a proton pump inhibitor at a stable dose.
* Patients with any other factor likely to alter intra-gastric acidity e.g. previous gastric surgery, including vagotomy or anatomically abnormal upper gastrointestinal tract.
* History of other malignant disease within the previous five years, except non- melanomatous skin cancer or in situ carcinoma of the uterine cervix.
* Previous use within the last four weeks, concomitant use or anticipated use in the period of the study of radiotherapy or chemotherapy.
* Concomitant use of immunosuppressants, including systemic (i .e. oral or injected) corticosteroids.
* Females who were pregnant, planning to become pregnant or lactating. Women, who in the opinion of the investigator were of child bearing potential, were to have a negative pregnancy test before study drug administration.
* Patients taking part in another study involving an investigational or licensed drug or device in the three months preceding enrolment or during the study.
* Previous G 17DT treatment.
* Haematological indicators:

Haemoglobin <10.0 g/dL White blood cell count <4.0 x 109/L Platelets < 100 x 1 09/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2001-08 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Antibody Levels | 12 weeks
  Assess effects of gastrin-17 antibodies in response to G17DT immunization.

SECONDARY OUTCOMES:
pharmacodynamic | 12 weeks
  measure production of gastrin-17 antibodies.
Number of Participants with Serious and Non-Serious Adverse Events | 12 weeks
  Adverse events, defined as any event involving adverse reactions, illnesses with onset during the study, or exacerbations of pre-existing illnesses, were assessed at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aintree, Liverpool, Merseyside, United Kingdom